CLINICAL TRIAL: NCT02960763
Title: Optimizing Outcomes of Treatment-Resistant Depression in Older Adults
Acronym: OPTIMUM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Eric Lenze, Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201609085; TRD-1511-33321 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2016-10-28; First posted 2016-11-10 (Estimated); Results first posted 2022-05-24 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Treatment Resistant Depression; Major Depressive Disorder; Treatment-Refractory Depression; Late Life Depression; Geriatric Depression
Keywords: Comparative Effectiveness Research; Pragmatic Clinical Trials; Patient-Centered Outcomes Research
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Aripiprazole; Bupropion; Lithium Carbonate; Nortriptyline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Aripiprazole Augmentation (Experimental): Augment current antidepressant treatment with aripiprazole (tablets), titrated from 2-15 mg daily based on symptom severity and side effects.
  Interventions: Drug: Aripiprazole Augmentation
- Bupropion Augmentation (Experimental): Augment current antidepressant treatment with bupropion once-daily extended release, titrated from 150-300 mg daily based on symptom severity and side effects.
  Interventions: Drug: Bupropion Augmentation
- Switch to Bupropion (Experimental): Taper from current antidepressant therapy. Start bupropion once-daily extended, titrated from 150-300 mg daily based on symptom severity and side effects.
  Interventions: Drug: Switch to bupropion
- Lithium Augmentation (Experimental): Augment current antidepressant treatment with lithium carbonate tablets starting at 300 mg daily, titrated per blood level to 0.4-0.6 meQ/L.
  Interventions: Drug: Lithium Augmentation
- Switch to Nortriptyline (Experimental): Taper from current antidepressant therapy. Start on nortriptyline tablets starting at 1 mg per kg of body weight daily, titrated per blood level to 80-120 ng/ml.
  Interventions: Drug: Switch to nortriptyline

INTERVENTIONS:
Drug: Aripiprazole Augmentation — Augment current antidepressant treatment with aripiprazole (tablets). Start at 2 mg daily; increase every two weeks (i.e., to 5, 7, 10 mg) to a maximum of 15 mg daily based on symptom severity and side effects.
  Other Names: Abilify
  Arms: Aripiprazole Augmentation
Drug: Bupropion Augmentation — Augment current antidepressant treatment with bupropion once-daily extended release, starting at 150 mg daily; titrated after four weeks to 300 mg daily based on symptom severity and side effects.
  Other Names: Wellbutrin
  Arms: Bupropion Augmentation
Drug: Switch to bupropion — Taper from current antidepressant therapy. Start bupropion once-daily extended release at 150 mg daily; titrated after four weeks to 300 mg daily based on symptom severity and side effects.
  Other Names: Wellbutrin
  Arms: Switch to Bupropion
Drug: Lithium Augmentation — Augment current antidepressant treatment with lithium carbonate tablets starting at 300 mg daily, titrated per blood level to 0.4-0.6 meQ/L.
  Other Names: Lithium carbonate; Eskalith
  Arms: Lithium Augmentation
Drug: Switch to nortriptyline — Taper from current antidepressant therapy. Start on nortriptyline tablets starting at 1 mg per kg of body weight daily, titrated per blood level to 80-120 ng/ml
  Other Names: Pamelor,
  Arms: Switch to Nortriptyline

SUMMARY:
The purpose of this research study is to assess which antidepressants work the best in older adults who have treatment-resistant depression (TRD).

DETAILED DESCRIPTION:
Older adult participants with treatment-resistant depression will be randomly assigned to a Step 1 medication strategy.

* Adding aripiprazole to current antidepressant medication
* Adding bupropion to current antidepressant medication
* Replacing current antidepressant medication with bupropion

If depression is not relieved at the end of 10 weeks, or if participants do not qualify for Step 1, participants will be randomly assigned to a Step 2 medication strategy:

* Adding lithium to current antidepressant medication
* Replacing current antidepressant medication with nortriptyline

All medication strategies will be offered in collaboration with participants' own physicians with the the research team providing support and guidance.

After treatment in Step 1 and/or Step 2, participants will enter the Continuation Phase to assess long term follow-up outcomes for 12 months.

Participants in this clinical trial will also be asked to participate in an additional study to gather imaging and biomarker data.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 60 and older
* Current Major Depressive Disorder (MDD)
* Failure to respond adequately to two or more antidepressant treatment trials of recommended dose and length
* Patient Health Questionnaire-9 (PHQ-9) score of 10 or higher

Exclusion Criteria:

* Inability to provide informed consent
* Dementia
* Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
* High risk for suicide and unable to be managed safely in the clinical trial
* Contraindication to proposed study medications, as determined by study physician including history of intolerance or non-response to proposed medications.
* Non-correctable, clinically significant sensory impairment interfering with participation
* Unstable medical illness, including delirium, uncontrolled diabetes mellitus, hypertension, hyperlipidemia, or cerebrovascular or cardiovascular risk factors that are not under medical management.
* Moderate to severe substance or alcohol use disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 742 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (5):
- United States (4):
  - UCLA Late-Life Mood, Stress, and Wellness Research Program, Los Angeles, California
  - Washington University School of Medicine Healthy Mind Lab, St Louis, Missouri
  - Columbia University Adult and Late Life Depression Clinic, New York, New York
  - UPMC Late-Life Depression, Evaluation, Prevention, and Treatment Program, Pittsburgh, Pennsylvania
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
A cleaned, complete, and de-identified copy of the final data set including administrative and technical metadata records will be made available through a Washington University in St. Louis (WUSTL) secure repository and registered at clinicaltrials.gov.

REFERENCES:
- [Derived] Oughli HA, Ainsworth NJ, Butters MA, Brown PJ, Gebara MA, Gettinger TR, Karp JF, Lavretsky H, Lenard E, Miller JP, Mulsant BH, Nicol GE, Reynolds CF 3rd, Yingling M, Lenze EJ; OPTIMUM Research Group. Cognitive changes in older adults receiving pharmacotherapy for treatment-resistant depression: a secondary analysis of the OPTIMUM randomised controlled trial. Lancet Healthy Longev. 2025 Oct;6(10):100767. doi: 10.1016/j.lanhl.2025.100767. Epub 2025 Nov 11. PMID 41237789
- [Derived] Srifuengfung M, Lenze EJ, Roose SP, Brown PJ, Lavretsky H, Karp JF, Reynolds CF 3rd, Yingling M, Sa-Nguanpanich N, Mulsant BH. Alcohol and substance use in older adults with treatment-resistant depression. Int J Geriatr Psychiatry. 2024 Jun;39(6):e6105. doi: 10.1002/gps.6105. PMID 38822571
- [Derived] Lenze EJ, Mulsant BH, Roose SP, Lavretsky H, Reynolds CF 3rd, Blumberger DM, Brown PJ, Cristancho P, Flint AJ, Gebara MA, Gettinger TR, Lenard E, Miller JP, Nicol GE, Oughli HA, Pham VT, Rollman BL, Yang L, Karp JF. Antidepressant Augmentation versus Switch in Treatment-Resistant Geriatric Depression. N Engl J Med. 2023 Mar 23;388(12):1067-1079. doi: 10.1056/NEJMoa2204462. Epub 2023 Mar 3. PMID 36867173

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited based on referrals from primary care providers (PCPs) or psychiatrists and self-referrals. This was further checked by using tools electronic medical records (EMRs) and using EMR-launched clinical decision tools. Print, radio, and social media advertising were used too. If patients self-referred, treatment recommendations were given by their community providers or a psychiatrist associated with the study.
Period: Step 1
Arm/Group | Aripiprazole Augmentation | Bupropion Augmentation | Switch to Bupropion | Lithium Augmentation | Switch to Nortriptyline
Started | 211 | 206 | 202 | 0 | 0
Completed ("Step 1" only includes: Aripiprazole Augmentation Bupropion Augmentation Switch to Bupropion) | 192 | 188 | 174 | 0 | 0
Not Completed | 19 | 18 | 28 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 8 | 13 | 0 | 0
Not completed — Lost to Follow-up | 7 | 9 | 12 | 0 | 0
Not completed — Death | 1 | 1 | 1 | 0 | 0
Not completed — Investigator discretion | 1 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Period: Step 2
Arm/Group | Aripiprazole Augmentation | Bupropion Augmentation | Switch to Bupropion | Lithium Augmentation | Switch to Nortriptyline
Started | 0 | 0 | 0 | 127 | 121
People Who Participated in Step 1 and Continued to Participate in Step 2 | 43 | 44 | 38 | 0 | 0
People Who Began Step 2 Without Having Participated in Step 1 | 0 | 0 | 0 | 63 | 60
Completed ("Step 2" only includes: Lithium Augmentation Switch to Nortriptyline) | 0 | 0 | 0 | 116 | 116
Not Completed | 0 | 0 | 0 | 11 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 7 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4 | 1
Not completed — Investigator discretion | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: In Participant Flow, Step 2 "milestones" shows numbers recorded for those who switched from Step 1 to Step 2, and the numbers for those who started Step 2 without having first participated in Step 1.
  125 participants from the Step 1 arms (aripiprazole augmentation, bupropion augmentation, and switch to bupropion) also participated in Step 2.
  A grand total of 742 unique participants were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole Augmentation | Bupropion Augmentation | Switch to Bupropion | Lithium Augmentation | Switch to Nortriptyline | Total
Number analyzed (Participants) | 211 | 206 | 202 | 127 | 121 | 867
Age, Continuous [Mean (Standard Deviation); unit: years] — Age for Step 1 participants Population: Step 1 had 619 participants enrolled
  years
    number analyzed (Participants) | 211 | 206 | 202 | 0 | 0 | 619
    (all) | 69.07 (6.46) | 69.13 (7.14) | 69.68 (7.71) |  |  | 69.29 (7.10)
Age, Customized [Mean (Standard Deviation); unit: years] — Age of Step 2 participants Population: Step 2 had 248 participants enrolled
  years
    number analyzed (Participants) | 0 | 0 | 0 | 127 | 121 | 248
    (all) |  |  |  | 69.04 (6.00) | 68.03 (5.72) | 68.55 (5.88)
Sex: Female, Male [Count of Participants; unit: Participants] — Step 1 participants Population: Step 1 totals for sex of participants enrolled
  Participants
    number analyzed (Participants) | 211 | 206 | 202 | 0 | 0 | 619
    Female | 144 | 142 | 127 |  |  | 413
    Male | 67 | 64 | 75 |  |  | 206
Sex: Female, Male [Count of Participants; unit: Participants] — Step 2 participants Population: Step 2 sex of participants enrolled
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 127 | 121 | 248
    Female |  |  |  | 90 | 83 | 173
    Male |  |  |  | 37 | 38 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Step 1 participants Population: Step 1 race/ethnicity of participants enrolled
  Participants
    White: number analyzed (Participants) | 211 | 206 | 202 | 0 | 0 | 619
    White | 173 | 174 | 175 |  |  | 522
    African American: number analyzed (Participants) | 211 | 206 | 202 | 0 | 0 | 619
    African American | 16 | 17 | 13 |  |  | 46
    Other: number analyzed (Participants) | 211 | 206 | 202 | 0 | 0 | 619
    Other | 22 | 15 | 14 |  |  | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Step 1 participants Population: Step 1 race/ethnicity of participants enrolled
  Participants
    Hispanic/Latino: number analyzed (Participants) | 211 | 206 | 202 | 0 | 0 | 619
    Hispanic/Latino | 22 | 17 | 13 |  |  | 52
    Other: number analyzed (Participants) | 211 | 206 | 202 | 0 | 0 | 619
    Other | 189 | 189 | 189 |  |  | 567
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Step 2 participants Population: Step 2 race/ethnicity of participants enrolled
  Participants
    White: number analyzed (Participants) | 0 | 0 | 0 | 127 | 121 | 248
    White |  |  |  | 116 | 106 | 222
    African American: number analyzed (Participants) | 0 | 0 | 0 | 127 | 121 | 248
    African American |  |  |  | 7 | 4 | 11
    Other: number analyzed (Participants) | 0 | 0 | 0 | 127 | 121 | 248
    Other |  |  |  | 4 | 11 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Step 2 participants Population: Step 2 race/ethnicity of participants enrolled
  Participants
    Hispanic/Latino: number analyzed (Participants) | 0 | 0 | 0 | 127 | 121 | 248
    Hispanic/Latino |  |  |  | 3 | 10 | 13
    Other: number analyzed (Participants) | 0 | 0 | 0 | 127 | 121 | 248
    Other |  |  |  | 124 | 111 | 235

OUTCOME MEASURES:

1. Primary Outcome: Psychological Well-Being
Description: Psychological well-being was assessed using the NIH Toolbox Psychological Wellbeing subscales of Positive Affect and General Life Satisfaction, with a T score calculated as the average of these two subscales. Higher scores indicate greater positive affect and life satisfaction. Reference T-score (mean=50, SD=10).
Time Frame: Step 1 (10 weeks), Step 2 (10 weeks), a period of up to 20 weeks
Measure: Mean (95% Confidence Interval); unit: t-score
Arm/Group | Aripiprazole Augmentation | Bupropion Augmentation | Switch to Bupropion | Lithium Augmentation | Switch to Nortriptyline
Number analyzed (Participants) | 211 | 206 | 202 | 127 | 121
t-score
  baseline | 34.7 [33.8 to 35.6] | 35.0 [34.1 to 36.0] | 34.8 [33.8 to 35.7] | 33.1 [31.9 to 34.4] | 34.2 [32.9 to 35.4]
  10 weeks | 38.8 [37.9 to 39.8] | 38.7 [37.8 to 39.7] | 36.1 [35.1 to 37.2] | 35.7 [34.4 to 37.1] | 35.6 [34.3 to 37.0]
Statistical Analysis 1: Comparison: Aripiprazole Augmentation vs Bupropion Augmentation vs Switch to Bupropion; Test type: Superiority — Repeated measure of 2*2*3 ANOVA with age (60 - 70, > 70), time (baseline, end of Active phase of Step 1) by treatment group (3 levels). Tests were conducted with a Hochberg Step-down procedure. If the comparison with the lowest p-value < 0.05/3 it is significant. If the second lowest p-value is also < 0.05/2 then it also will be significant and if the third p-value is < 0.05 then it also will be significant; p = 0.010, ANOVA — Equivalence of group
Statistical Analysis 2: Comparison: Aripiprazole Augmentation vs Switch to Bupropion; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.004, ANOVA — augment with aripiprazole vs switch to bupropion
Statistical Analysis 3: Comparison: Bupropion Augmentation vs Switch to Bupropion; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.017, ANOVA — augment with bupropion vs switch to bupropion
Statistical Analysis 4: Comparison: Aripiprazole Augmentation vs Bupropion Augmentation; Repeated measure of 2*2*3 ANOVA with age (60 - 70, > 70), time (baseline, end of Active phase of Step 1) by treatment group (3 levels). Tests were conducted with a Hochberg Step-down procedure. If the comparison with the lowest p-value < 0.05/3 it is significant. If the second lowest p-value is also < 0.05/2 then it also will be significant and if the third p-value is < 0.05 then it also will be significant; Test type: Superiority; p = 0.650, ANOVA
Statistical Analysis 5: Comparison: Aripiprazole Augmentation vs Bupropion Augmentation vs Switch to Bupropion; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.003, ANOVA — augmentation versus switch
Statistical Analysis 6: Comparison: Lithium Augmentation vs Switch to Nortriptyline; Test type: Superiority — For those who proceed to Step 2, analogous repeated measures 2*2*2 ANOVA will be used with a significance level of .05 for the time*treatment group comparison; p = 0.385, ANOVA

2. Primary Outcome: Number of Participants With Remission From Depression
Description: Remission defined as Montgomery Asberg Depression Rating Scale score ≤10. Scale ranges from 0-60 with higher scores indicating higher depressive symptoms.
Time Frame: Step 1 (10 weeks), Step 2 (10 weeks), a period of up to 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole Augmentation | Bupropion Augmentation | Switch to Bupropion | Lithium Augmentation | Switch to Nortriptyline
Number analyzed (Participants) | 211 | 206 | 202 | 127 | 121
Participants | 61 | 58 | 39 | 24 | 26
Statistical Analysis 1: Comparison: Aripiprazole Augmentation vs Bupropion Augmentation vs Switch to Bupropion; Test type: Superiority; p = 0.038, generalized linear model with logistic l — Group effect
Statistical Analysis 2: Comparison: Aripiprazole Augmentation vs Switch to Bupropion; Test type: Superiority; p = 0.021, generalized linear model with logistic l — augmentation with aripiprazole vs switch to bupropion
Statistical Analysis 3: Comparison: Bupropion Augmentation vs Switch to Bupropion; Test type: Superiority; p = 0.027, generalized linear model with logistic l — augmentation with bupropion vs switch to bupropion
Statistical Analysis 4: Comparison: Aripiprazole Augmentation vs Bupropion Augmentation; Test type: Superiority; p = 0.934, generalized linear model with logistic l — Augmentation with aripiprazole v augmentation with bupropion
Statistical Analysis 5: Comparison: Aripiprazole Augmentation vs Bupropion Augmentation vs Switch to Bupropion; Test type: Superiority; p = 0.011, generalized linear model with logistic l — augmentation versus switch
Statistical Analysis 6: Comparison: Lithium Augmentation vs Switch to Nortriptyline; Test type: Superiority; p = 0.500, generalized linear model with logistic l

3. Primary Outcome: Serious Adverse Events
Description: Life threatening illness, hospitalization, or need of medical care.
Time Frame: Step 1 (10 weeks), Step 2 (10 weeks), a period of up to 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Aripiprazole Augmentation | Bupropion Augmentation | Switch to Bupropion | Lithium Augmentation | Switch to Nortriptyline
Number analyzed (Participants) | 211 | 206 | 202 | 127 | 121
Participants | 15 | 15 | 19 | 12 | 11
Statistical Analysis 1: Comparison: Aripiprazole Augmentation vs Bupropion Augmentation vs Switch to Bupropion; Test type: Superiority; p = 0.164, Regression, Cox — Cox models time to event comparing treatment arms
Statistical Analysis 2: Comparison: Aripiprazole Augmentation vs Switch to Bupropion; Test type: Superiority; p = 0.103, Regression, Cox
Statistical Analysis 3: Comparison: Bupropion Augmentation vs Switch to Bupropion; Test type: Superiority; p = 0.127, Regression, Cox
Statistical Analysis 4: Comparison: Lithium Augmentation vs Switch to Nortriptyline; Test type: Superiority; p = 0.524, Regression, Cox — Cox models to examine time to event comparing treatment arms

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during phone assessments every other week during Step 1 and Step 2 (approximately 10 weeks each) for approximately 20 weeks of event data.
Description: This study assessed adverse events (in particular falls) to determine how safe and tolerable the treatments were. This was done because it is important for doctors to be able to cite safety concerns as one of the main restrictions in treatment of depression in older adults. One challenge with the rates of AE's/SAE's was because of the naturally high rate of medical problems and falls in depressed older adults. Most of the SAE's reported were decided to not be related to treatment.
Arm/Group | Aripiprazole Augmentation | Bupropion Augmentation | Switch to Bupropion | Lithium Augmentation | Switch to Nortriptyline
All-Cause Mortality (participants affected / at risk) | 1/211 | 1/206 | 1/202 | 0/127 | 0/121
Serious Adverse Events (participants affected / at risk) | 15/211 | 15/206 | 19/202 | 12/127 | 11/121
Other Adverse Events (participants affected / at risk) | 148/211 | 120/206 | 136/202 | 93/127 | 93/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole Augmentation (N=211) | Bupropion Augmentation (N=206) | Switch to Bupropion (N=202) | Lithium Augmentation (N=127) | Switch to Nortriptyline (N=121)
Psychiatric Hospitalization (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Non-psychiatric Hospitalization (General disorders) | 14 (14) | 11 (11) | 17 (22) | 12 (13) | 8 (8)
Fall (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — required surgery/ER visit, but no known overnight hospitalization
Other (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — includes instances of unrelated cancer and death to unrelated study cause
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole Augmentation (N=211) | Bupropion Augmentation (N=206) | Switch to Bupropion (N=202) | Lithium Augmentation (N=127) | Switch to Nortriptyline (N=121)
Akathisia (Psychiatric disorders) | 23 | 2 | 5 | 2 | 0 — Unable to be still, and having the constant urge to move
Headache (General disorders) | 16 | 17 | 15 | 13 | 6
Reduced Salivation (General disorders) | 15 | 30 | 23 | 13 | 51 — dryness of mouth
Nausea/Vomiting (Gastrointestinal disorders) | 15 | 25 | 31 | 12 | 9
Diarrhea (Gastrointestinal disorders) | 14 | 12 | 11 | 8 | 7
Constipation (Gastrointestinal disorders) | 15 | 20 | 18 | 6 | 20
Weight gain (General disorders) | 32 | 3 | 1 | 8 | 4
Cold/Flu Symptoms (General disorders) | 29 | 18 | 23 | 13 | 13
Dizziness (General disorders) | 36 | 41 | 40 | 28 | 21
Fall (General disorders) | 11 | 16 | 15 | 10 | 5
Increased Appetite Without Weight Gain (General disorders) | 23 | 2 | 6 | 2 | 6
Irritability or Emotional Lability (Psychiatric disorders) | 10 | 12 | 34 | 5 | 15
Concenctration Difficulties (Psychiatric disorders) | 11 | 4 | 10 | 9 | 10
Asthenia/Lassitude/Increased Fatiguability (General disorders) | 18 | 11 | 3 | 18 | 11
Sleepiness/Sedation (General disorders) | 20 | 9 | 3 | 11 | 12
Tension/Inner Unrest (General disorders) | 30 | 20 | 29 | 8 | 9
Tremor (General disorders) | 14 | 20 | 13 | 34 | 4
Polyuria/Polydipsia (Renal and urinary disorders) | 5 | 0 | 6 | 11 | 1 — frequent need to urinate/feeling of extreme thirstiness
Increased Tendency to Sweating (General disorders) | 5 | 8 | 5 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT02960763/Prot_002.pdf
  • Statistical Analysis Plan (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT02960763/SAP_004.pdf